CLINICAL TRIAL: NCT03784222
Title: Effects on Social and Cognition Functions of Blonanserin in First Episode Schizophrenia Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Company's business decision
Sponsor: Sumitomo Pharma (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSPCLON-002
Record Dates: First submitted 2018-11-28; First posted 2018-12-21 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: First Episode Schizophrenia; Social Function; Cognition Function; Blonanserin
MeSH Terms: conditions — Social Adjustment | interventions — blonanserin; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): 188 first episode schizophrenia patients, receiving blonanserin treatment, 60 of the patients receive MRI and serum BDNF test
  Interventions: Drug: Blonanserin; Other: MRI and serum BDNF
- control group (Other): 60 subjects without schizophrenia, only receiving MRI and/or serum BDNF
  Interventions: Other: MRI and serum BDNF

INTERVENTIONS:
Drug: Blonanserin — patients were prescribed blonanserin 4-24mg/d according to the patients' response and tolerability
  Arms: treatment group
Other: MRI and serum BDNF — 60 patients receive MRI and serum BDNF test, 60 controls receive MRI, 20 of the 60 controls receive serum BDNF test

SUMMARY:
This is an open label, multi-center study to explore the effects on social functions of blonanserin in first episode schizophrenia patients

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia patients diagnosis either with DSM-5 criteria or ICD-10;
* PANSS total score ≥70;
* Males or Females aged 18-45 years;
* With disease course less than 5 years and during their first episode;
* ≥9 years of education;
* Without receiving systematic antipsychotic treatment, or receiving continuous antipsychotic treatment for less than 6 weeks and receiving antipsychotic treatment for less than 6 months in total;
* Ability to read and understand Chinese;
* Provision of written informed consent

Exclusion Criteria:

* Severe or unstable physical diseases judged by investigators;
* Loss of consciousness more than 1 hour due to any reason in the past 1 year;
* Current substance misuse (in 3 months) or any substance dependence;
* Pregnant or lactating woman;
* Patients with attempted suicide history, severe suicidal ideation or behaviour;
* Mental retardation;
* Contradict to the study drugs;
* Patients taken other investigation products in the past 30 days before entry;
* Patients ever taken blonanserin before;
* Any current medical condition that would interfere with the assessment of efficacy;
* Physical symptoms of acute deterioration requiring hospitalization or increased intensive care;
* Significant muscle tension or Parkinson's disease;
* Clinically significant abnormal laboratory test results (blood, urine, and blood biochemical analysis);
* Clinically significant Abnormal electrocardiogram as judged by researchers;
* Participants continuously using sedative drugs, or anticholinergic agents within 3 months of the study;
* Those who had undergone electroconvulsive therapy within 3 month of the study;
* Those who had received long-acting injection treatment within 3 month of the study;
* Those who could not swallow medication with water;
* Subjects judged by the investigator in charge as inappropriate for the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
changes in personal and social performance (PSP) scores at week 26 | 26 weeks
  PSP consists of four main areas: 1. Socially useful activities (e.g., housework, voluntary work) including work and study; 2. Personal and social relationships (i.e., partner, family relationships, friends); 3. Self-care (i.e., personal hygiene, care of one's appearance); 4. Disturbing and aggressive behavior. The maximum scores is 100, the minimum scores is 1, higher values represent a better outcome

SECONDARY OUTCOMES:
changes in MATRICS Consensus Cognitive Battery (MCCB) domain scores at week 26 in treatment group | 26 weeks
  MATRICS Consensus Cognitive Battery (MCCB) includes 10 tests that measure seven cognitive domains: speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving and social cognition. Scores for the individual tests will be calculated according to the developer's recommended scoring algorithms
changes in Paced Auditory Serial Addition Task (PASAT) test at week 26 in treatment group | 26 weeks
  PASAT is a neuropsychological test used to assess capacity and rate of information processing and sustained and divided attention
changes in Groove Pegboard Test (GPT) at week 26 in treatment group | 26 weeks
  GPT is a test used to assess fine motor skills and speed. this test measure the time it takes to put 25 nails in the pegborad in a defined order
changes in positive and negative syndrome scale (PANSS) total scores at week 26 in treatment group | 26 weeks
  PANSS is a medical scale used for measuring symptom severity of patients with schizophrenia. the maximum scores is 210, the minimum scores is 30. the higher values represent a worse outcome. the total scores are the sum of subscales.
changes in PANSS five-factor model scores at week 26 in treatment group | 26 weeks
  five-factor model is another model of PANSS. It is a medical scale used for measuring symptom severity of patients with schizophrenia. the maximum scores is 210, the minimum scores is 30. the higher values represent a worse outcome. the total scores are the sum of subscales.
changes in PSP at every visit in treatment group during 26 weeks | baseline, week 8, week 26
  PSP consists of four main areas: 1. Socially useful activities (e.g., housework, voluntary work) including work and study; 2. Personal and social relationships (i.e., partner, family relationships, friends); 3. Self-care (i.e., personal hygiene, care of one's appearance); 4. Disturbing and aggressive behavior. The maximum scores is 100, the minimum scores is 1, higher values represent a better outcome
changes in MCCB at every visit in treatment group during 26 weeks | baseline, week 8, week 26
  MATRICS Consensus Cognitive Battery (MCCB) includes 10 tests that measure seven cognitive domains: speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving and social cognition. Scores for the individual tests will be calculated according to the developer's recommended scoring algorithms

OTHER OUTCOMES:
changes in magnetic resonance imaging (MRI) at week 26 in treatment group | 26 weeks
  observe the change of grey matter volume, white matter volume, and the functions and connections in different encephalic regions
changes in MRI at every visit in treatment group during 26 weeks | baseline, week 8, week 26
  observe the change of grey matter volume, white matter volume, and the functions and connections in different encephalic regions
difference of MRI results between treatment group and control group at baseline | baseline
  observe the change of grey matter volume, white matter volume, and the functions and connections in different encephalic regions
changes in serum Brain-derived neurotrophic factor (BDNF) at week 26 in treatment group | 26 weeks
  BDNF, is a protein that, in humans, is encoded by the BDNF gene. BDNF is a member of the neurotrophin family of growth factors, which are related to the canonical nerve growth factor. Neurotrophic factors are found in the brain and the periphery
difference of serum BDNF results between treatment group and control group at baseline | baseline
  BDNF, is a protein that, in humans, is encoded by the BDNF gene. BDNF is a member of the neurotrophin family of growth factors, which are related to the canonical nerve growth factor. Neurotrophic factors are found in the brain and the periphery

CONTACTS AND LOCATIONS:
Overall Officials: Xin Yu, MD, Principal Investigator — Peking University Sixth Hospital
Locations (8):
- China (8):
  - Beijing Huilongguan Hospital, Beijing, Beijing Municipality
  - Peking University Sixth Hospital, Beijing, Beijing Municipality
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - Xi'an Mental Health Center, Xi’an, Shanxi
  - West China Hospital, Sichuan Univeristy, Chengdu, Sichuan
  - Tianjin Mental Health Center, Tianjin, Tianjin Municipality
  - The First Affiliated hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pu C, Lei L, Yang F, Deng H, Sheng J, Liu Z, Hu S, Wang L, Wu B, Bo Q, Inoue Y, Yu X. Effectiveness and safety of blonanserin for improving social and cognitive functions in patients with first-episode schizophrenia: a study protocol for a prospective, multicentre, single-arm clinical trial. BMJ Open. 2022 Apr 20;12(4):e054079. doi: 10.1136/bmjopen-2021-054079. PMID 35443947